CLINICAL TRIAL: NCT05712252
Title: Risk Factors for Fall and Fracture - A Cohort Study of Fall-related Factors Obtained in Routine Orthopaedic Fracture Care
Brief Title: Fall, Fracture and Frailty
Acronym: FFF
Status: Active, not recruiting | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-01997-01
Record Dates: First submitted 2023-01-11; First posted 2023-02-03 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Fall Injury; Hip Fractures; Risk Reduction; Osteoporosis, Osteopenia; Frailty
Keywords: Falls; Fracture; Frailty; Orthogeriatric
MeSH Terms: conditions — Hip Fractures; Risk Reduction Behavior; Osteoporosis; Bone Diseases, Metabolic; Frailty; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fallers without a fracture: Individuals who obtain no fracture.
- Fallers with a fracture: Individuals who obtain one or several fractures through fall. This group can be further subgrouped according to type of fracture.

SUMMARY:
This project aims to improve the global outcome for an aging individual after a traumatic fall, through identifying conditions contributing to a fall and promoting recovery and rehabilitation. Through better understanding 'falling phenotype', the ultimate aim is to prevent future complications, as well as new falls and fractures in the growing older population.

DETAILED DESCRIPTION:
Background: The knowledge of risk factors for falls and fractures amongst older individuals are enormous, still identification of fallers and prevention of falls is not part of Swedish standard of care. Some risk factors are more or less overlooked, such as alcohol consumption, orthostatic reactions, as are increased risks related to common medications such as certain antidepressants, opioids and sedatives. Although functional activity and frailty scores have been suggested to be potential predictors of adverse events, length of hospital stay and mortality, the use of standardized questionnaires has not been implemented in routine care in Sweden. Furthermore, outcomes after fragility fractures, a well known consequence of falls among older individuals, are continuously poor, although palpable improvements have been reached regarding surgical treatment. Are there other factors that are equally or more decisive for the global outcome from the patient's point of view?

Material & Methods: In this prospective observational cohort study, all in-patients treated due to a fall-related trauma (fracture, dislocation or contusion) at the Department of Orthopaedics, Skane University Hospital Malmö, aged 65 years or older will be invited to participate during a 1-year study period. In all participants, a standard package of blood samples, temperature, measurement of orthostatic blood pressure and grip strength, grading of frailty and activity will be routinely obtained.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older at the time of admission.
* Admitted to Orthopaedic ward at due to fall, with or without a fracture.

Exclusion Criteria:

* Severe head trauma or other severe non-orthopaedic trauma.
* Other condition requiring ward at other department (CCU, ICU) >24 hours.
* Moribund individuals with palliative care only.
* Declined to participate
* Fall > 7 days before admission
* Residence outside the region (lack of follow-up)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Individuals aged 65 years or older who are admitted to Orthopaedic ward at Skåne University Hospital in Malmö, due to a fall or fall-related trauma.
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-10-06 (Actual); Study Completion 2027-09-06 (Estimated)

PRIMARY OUTCOMES:
Mortality | One year after admission to hospital
  The number of deaths during follow-up
Re-admission | One year after admission to hospital
  Number of re-admissions to emergency centre or in-patient ward due to a new fall (primarily) or complications related previous fall/fracture
Other adverse events | One year after admission to hospital
  Other adverse events that are not included in outcome measure 1 or 2, such as infection, new falls, fractures, or complications from previous fall/fracture, or other medical complications. These can be further grouped by whether the events occur in in-patient or out-patient care.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Rogmark, MD, PhD, Principal Investigator — Department of Orthopaedics, Skåne University Hospital, Malmö, Sweden
Locations (1):
- Department of Orthopaedics, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual participant data are not publicly available because of patient integrity but anonymized, supplementary data supporting the findings of individual studies are available upon reasonable request to the corresponding author.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-13): https://cdn.clinicaltrials.gov/large-docs/52/NCT05712252/Prot_SAP_001.pdf